CLINICAL TRIAL: NCT01497899
Title: A Phase 2, Randomized, Double-Blinded Study of the Safety and Efficacy of Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide Single Tablet Regimen Versus Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Disoproxil Fumarate Single Tablet Regimen in HIV-1 Infected, Antiretroviral Treatment-Naive Adults
Brief Title: Safety and Efficacy of E/C/F/TAF (Genvoya®) Versus E/C/F/TDF (Stribild®) in HIV-1 Infected, Antiretroviral Treatment-Naive Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-292-0102
Record Dates: First submitted 2011-12-14; First posted 2011-12-23 (Estimated); Results first posted 2016-01-08 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2017-08

CONDITIONS: Acquired Immunodeficiency Syndrome; HIV Infections
Keywords: HIV-1; HIV; Treatment-Naive
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- E/C/F/TAF (Experimental): E/C/F/TAF plus E/C/F/TDF placebo for at least 48 weeks
  Interventions: Drug: E/C/F/TAF; Drug: E/C/F/TDF Placebo
- E/C/F/TDF (Active Comparator): E/C/F/TDF plus E/C/F/TAF placebo for at least 48 weeks
  Interventions: Drug: E/C/F/TDF; Drug: E/C/F/TAF Placebo
- E/C/F/TAF Open-Label (Experimental): Following study unblinding, participants from the E/C/F/TAF and E/C/F/TDF arms may have the option to receive E/C/F/TAF during an open-label extension phase.
  Also, participants who are actively participating in a Gilead-sponsored study of cobicistat-boosted darunavir plus nucleoside/nucleotide reverse transcriptase inhibitors (NRTI) who have reached the protocol-defined secondary endpoint (Week 48) and remain virologically suppressed are eligible to participate and receive E/C/F/TAF in this open-label extension phase.
  Interventions: Drug: E/C/F/TAF

INTERVENTIONS:
Drug: E/C/F/TDF — 150/150/200/300 mg FDC tablet administered orally once daily
  Other Names: Stribild®
  Arms: E/C/F/TDF
Drug: E/C/F/TAF Placebo — Tablet administered orally once daily
  Arms: E/C/F/TDF
Drug: E/C/F/TAF — 150/150/200/10 mg FDC tablet administered orally once daily
  Other Names: Genvoya®
  Arms: E/C/F/TAF; E/C/F/TAF Open-Label
Drug: E/C/F/TDF Placebo — Tablet administered orally once daily
  Arms: E/C/F/TAF

SUMMARY:
The primary objective of this study is to evaluate the efficacy of elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (Genvoya®; E/C/F/TAF) fixed-dose combination (FDC) versus elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate (Stribild®; E/C/F/TDF) FDC in HIV-1 infected, antiretroviral treatment-naive adults.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability to understand and sign a written informed consent form
* Plasma HIV 1 RNA levels ≥ 5,000 copies/mL
* No prior use of any approved or experimental anti-HIV drug for any length of time
* Screening genotype report must show sensitivity to TDF and emtricitabine (FTC)
* Normal ECG
* Adequate renal function: Estimated glomerular filtration rate ≥ 70 mL/min according to the Cockcroft Gault formula
* Hepatic transaminases ≤ 2.5 x upper limit of the normal range (ULN)
* Total bilirubin ≤ 1.5 mg/dL, or normal direct bilirubin
* Adequate hematologic function
* CD4+ cell count > 50 cells/µL
* Serum amylase ≤ 5 x ULN
* Normal thyroid-stimulating hormone (TSH)
* Females of childbearing potential must have a negative serum pregnancy test
* Females of childbearing potential must agree to utilize highly effective contraception methods from screening throughout the duration of study treatment and for 30 days following the last dose of study drugs
* Female subjects who utilize hormonal contraceptive as one of their birth control methods must have used the same method for at least three months prior to study dosing
* Female subjects who are postmenopausal must have documentation of cessation of menses for ≥ 12 months and hormonal failure
* Female subjects who have stopped menstruating for ≥ 12 months but do not have documentation of ovarian hormonal failure must have a serum follicle stimulating hormone (FSH) level test at screening
* Male subjects must agree to utilize a highly effective method of contraception during heterosexual intercourse throughout the study period and for 90 days following discontinuation of investigational medicinal product
* Age ≥ 18 years
* Life expectancy ≥ 1 year

Key Exclusion Criteria:

* New AIDS-defining condition diagnosed within the 30 days prior to screening
* Hepatitis B surface Antigen positive
* Hepatitis C Antibody positive
* Proven acute hepatitis in the 30 days prior to study entry
* Subjects experiencing decompensated cirrhosis
* Females who are breastfeeding
* Positive serum pregnancy test (female of childbearing potential)
* Have an implanted defibrillator or pacemaker
* Receiving ongoing therapy with any of the disallowed medications, including drugs not to be used with elvitegravir and cobicistat
* Have been treated with immunosuppressant therapies or chemotherapeutic agents within 3 months of study screening, or expected to receive these agents or systemic steroids during the study
* Current alcohol or substance
* History of or ongoing malignancy (including untreated carcinoma in-situ) other than cutaneous Kaposi's sarcoma (KS), basal cell carcinoma or resected, non-invasive cutaneous squamous carcinoma
* Active, serious infections (other than HIV 1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to Baseline
* Participation in any other clinical trial without prior approval is prohibited while participating in this trial
* Medications contraindicated for use with emtricitabine or tenofovir disoproxil fumarate
* Any known allergies to the excipients of E/C/F/TAF or E/C/F/TDF FDC tablets
* Any other clinical condition or prior therapy that would make the subject unsuitable for the study or unable to comply with the dosing requirements

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2011-12-28 (Actual); Primary Completion 2012-10-17 (Actual); Study Completion 2016-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (41):
- United States (40):
  - University of Alabama at Birmingham (UAB), Birmingham, Alabama
  - Spectrum Medical Group, Phoenix, Arizona
  - AHF Research Center, Beverly Hills, California
  - Kaiser Permanente, Los Angeles, California
  - Peter J. Ruane, MD, Inc., Los Angeles, California
  - Anthony Mills MD, Inc, Los Angeles, California
  - East Bay AIDS Center, Oakland, California
  - St. Joseph Heritage Healthcare, Orange, California
  - Stanford University, Palo Alto, California
  - Kaiser Permanente Medical Group, Sacramento, California
  - La Playa Medical Group and Clinical Research, San Diego, California
  - Metropolis Medical, San Francisco, California
  - Kaiser Permanente Medical Group-Clinical Trials Unit, San Francisco, California
  - Apex Research, LLC, Denver, Colorado
  - Dupont Circle Physician's Group, Washington D.C., District of Columbia
  - Whitman-Walker Health, Washington D.C., District of Columbia
  - Capital Medical Associates, PC, Washington D.C., District of Columbia
  - Gary J. Richmond,M.D.,P.A., Fort Lauderdale, Florida
  - Wohlfeiler, Piperato and Associates, LLC, Miami Beach, Florida
  - Orlando Immunology Center, Orlando, Florida
  - IDOCF/ValuhealthMD, LLC, Orlando, Florida
  - St. Joseph's Comprehensive Research Institute, Tampa, Florida
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Mercer University Mercer Medicine, Macon, Georgia
  - Howard Brown Health Center, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Be Well Medical Center, Berkley, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Central West Clinical Research Inc, St Louis, Missouri
  - North Shore University Hospital / Division of Infectious Diseases, Manhasset, New York
  - ID Consultants, P.A., Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of South Carolina School of Medicine Division of Infectious Disease, Columbia, South Carolina
  - Southwest Infectious Disease Clinical Research Inc, Dallas, Texas
  - Tarrant County Infectious Disease Associates, Fort Worth, Texas
  - Therapeutic Concepts, PA, Houston, Texas
  - Gordon E. Crofoot, MD., PA, Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Peter Shalit, M.D., Seattle, Washington
- Clinical Research Puerto Rico, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Sax PE, Zolopa A, Brar I, Elion R, Ortiz R, Post F, Wang H, Callebaut C, Martin H, Fordyce MW, McCallister S. Tenofovir alafenamide vs. tenofovir disoproxil fumarate in single tablet regimens for initial HIV-1 therapy: a randomized phase 2 study. J Acquir Immune Defic Syndr. 2014 Sep 1;67(1):52-8. doi: 10.1097/QAI.0000000000000225. PMID 24872136

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States and Puerto Rico. The first participant was screened on 28 December 2011. The last study visit occurred on 22 August 2016.
Pre-assignment Details: 232 participants were screened for the Double-Blind Phase. 108 participants from other Gilead-sponsored Study GS-US-299-0102 joined the Open-Label Extension Phase.
Groups:
- E/C/F/TAF: Double-Blind Phase: Elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (Genvoya®; E/C/F/TAF) (150/150/200/10 mg) fixed-dose combination (FDC) tablet plus elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate (Stribild®; E/C/F/TDF) placebo tablet administered orally once daily for 48 weeks
  Open-Label (OL) Extension Phase: E/C/F/TAF (150/150/200/10 mg) FDC tablet administered orally once daily
- E/C/F/TDF: Double-Blind Phase: E/C/F/TDF (150/150/200/300 mg) FDC tablet plus E/C/F/TAF placebo tablet administered orally once daily for 48 weeks
  Open-Label Extension Phase: E/C/F/TAF (150/150/200/10 mg) FDC tablet administered orally once daily
- D/C/F/TAF to Open-Label E/C/F/TAF: Participants previously received darunavir/cobicistat/emtricitabine/tenofovir alafenamide (D/C/F/TAF) in another Gilead-sponsored study and then enrolled into the Open-Label Extension Phase of this study to receive E/C/F/TAF (150/150/200/10 mg) FDC tablet administered orally once daily.
- DRV+COBI+TVD to Open-Label E/C/F/TAF: Participants previously received darunavir (DRV) + cobicistat (COBI) + Truvada® (TVD) in another Gilead-sponsored study and then enrolled into the Open-Label Extension Phase of this study to receive E/C/F/TAF (150/150/200/10 mg) FDC tablet administered orally once daily.
Period: Double-Blind Phase
Arm/Group | E/C/F/TAF | E/C/F/TDF | D/C/F/TAF to Open-Label E/C/F/TAF | DRV+COBI+TVD to Open-Label E/C/F/TAF
Started | 113 | 58 | 0 | 0
Completed | 107 | 53 | 0 | 0
Not Completed | 6 | 5 | 0 | 0
Not completed — Randomized but not Treated | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Investigator's Discretion | 1 | 0 | 0 | 0
Not completed — Withdrew Consent | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 3 | 2 | 0 | 0
Not completed — Subject Non-Compliance | 0 | 1 | 0 | 0
Period: Open-Label Extension Phase
Arm/Group | E/C/F/TAF | E/C/F/TDF | D/C/F/TAF to Open-Label E/C/F/TAF | DRV+COBI+TVD to Open-Label E/C/F/TAF
Started | 105 (2 participants completed the Double-Blind Phase, but did not continue in the Open-Label Extension.) | 53 | 70 (Participants enrolled from other Gilead-sponsored Study GS-US-299-0102.) | 38 (Participants enrolled from other Gilead-sponsored Study GS-US-299-0102.)
Completed | 86 | 46 | 61 | 33
Not Completed | 19 | 7 | 9 | 5
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Withdrew Consent | 8 | 3 | 2 | 0
Not completed — Pregnancy | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 9 | 3 | 5 | 5

BASELINE CHARACTERISTICS:
Population: E/C/F/TAF and E/C/F/TDF arms: participants who were randomized to the Double-Blind Phase and received at least 1 dose of study drug.
  D/C/F/TAF to E/C/F/TAF and DRV+COBI+TVD to E/C/F/TAF arms: participants who enrolled from Gilead-sponsored Study GS-US-299-0102 in the Open-Label Extension Phase and received at least 1 dose of open-label E/C/F/TAF
Groups:
- E/C/F/TAF: Double-Blind Phase: E/C/F/TAF (150/150/200/10 mg) FDC tablet plus E/C/F/TDF placebo tablet administered orally once daily for 48 weeks
  Open-Label (OL) Extension Phase: E/C/F/TAF (150/150/200/10 mg) FDC tablet administered orally once daily
- D/C/F/TAF to Open-Label E/C/F/TAF: Participants previously received D/C/F/TAF in another Gilead-sponsored study and then enrolled into the Open-Label Extension Phase of this study to receive E/C/F/TAF (150/150/200/10 mg) FDC tablet administered orally once daily.
- DRV+COBI+TVD to Open-Label E/C/F/TAF: Participants previously received DRV+COBI+TVD in another Gilead-sponsored study and then enrolled into the Open-Label Extension Phase of this study to receive E/C/F/TAF (150/150/200/10 mg) FDC tablet administered orally once daily.
- Total: Total of all reporting groups
Arm/Group | E/C/F/TAF | E/C/F/TDF | D/C/F/TAF to Open-Label E/C/F/TAF | DRV+COBI+TVD to Open-Label E/C/F/TAF | Total
Number analyzed (Participants) | 112 | 58 | 70 | 38 | 278
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (11.3) | 37 (10.6) | 36 (11.2) | 37 (10.7) | 36 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 3 | 3 | 11
  Male | 108 | 57 | 67 | 35 | 267

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 24
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 24 was analyzed using the snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 24
Population: Full Analysis Set: participants randomized to the Double-Blind Phase and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 112 | 58
percentage of participants | 88.4 | 89.7
Statistical Analysis 1: Comparison: E/C/F/TAF vs E/C/F/TDF; Test type: Non-Inferiority or Equivalence — The null hypothesis was that the E/C/F/TAF group was at least 12% lower than the E/C/F/TDF group with respect to the percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 24. The alternative hypothesis was that the E/C/F/TAF group was less than 12% lower than the E/C/F/TDF group; p = 0.58, Cochran-Mantel-Haenszel; P-value comparing the percentages of virologic success was from the Cochran-Mantel-Haenszel (CMH) test stratified by baseline HIV-1 RNA stratum; Difference in percentages = -2.9, 95% CI 2-sided [-13.5 to 7.7] — Difference in percentages of virologic success and its 95% confidence interval (CI) were calculated based on baseline HIV-1 RNA stratum-adjusted Mantel-Haenszel (MH) proportion

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 112 | 58
percentage of participants | 88.4 | 87.9

3. Secondary Outcome: Change From Baseline in log10 HIV-1 RNA at Weeks 24 and 48
Time Frame: Baseline; Weeks 24 and 48
Population: Participants in Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 112 | 58
log10 copies/mL
  Baseline | 4.63 (0.572) | 4.69 (0.577)
  Change at Week 24: number analyzed (Participants) | 108 | 58
  Change at Week 24 | -3.20 (0.654) | -3.26 (0.606)
  Change at Week 48: number analyzed (Participants) | 107 | 56
  Change at Week 48 | -3.22 (0.606) | -3.33 (0.572)

4. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Weeks 24 and 48
Time Frame: Baseline; Weeks 24 and 48
Population: Participants in Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 112 | 58
cells/uL
  Baseline | 404 (181.6) | 394 (209.6)
  Change at Week 24: number analyzed (Participants) | 108 | 58
  Change at Week 24 | 165 (115.6) | 179 (127.7)
  Change at Week 48: number analyzed (Participants) | 107 | 56
  Change at Week 48 | 177 (144.1) | 204 (120.4)

ADVERSE EVENTS:
Time Frame: Up to 186.2 weeks plus 30 days
Description: * Safety Analysis Set: participants who were enrolled and received at least 1 dose of study drug.
  * Double-blind phase (E/C/F/TAF and E/C/F/TDF arms): adverse events were coded using the Medical Dictionary for Regulated Activities (MedDRA), version 17.0
  * All E/C/F/TAF arm: adverse events were coded using MedDRA, version 19.0
Groups:
- E/C/F/TAF: Adverse events in this reporting group include those that occurred during the double-blind phase by participants randomized to E/C/F/TAF.
  Double-Blind Phase: E/C/F/TAF (150/150/200/10 mg) FDC tablet plus E/C/F/TDF placebo tablet administered orally once daily for 48 weeks; Open-Label (OL) Extension Phase: E/C/F/TAF (150/150/200/10 mg) FDC tablet administered orally once daily
- E/C/F/TDF: Adverse events in this reporting group include those that occurred during the double-blind phase by participants randomized to E/C/F/TDF.
  Double-Blind Phase: E/C/F/TDF (150/150/200/300 mg) FDC tablet plus E/C/F/TAF placebo tablet administered orally once daily for 48 weeks; Open-Label Extension Phase: E/C/F/TAF (150/150/200/10 mg) FDC tablet administered orally once daily
- All E/C/F/TAF: Adverse events in this reporting group include those that occurred any time during the study by participants while receiving E/C/F/TAF.
  Participants received blinded or open-label E/C/F/TAF (150/150/200/10 mg) FDC tablet administered orally once daily
Arm/Group | E/C/F/TAF | E/C/F/TDF | All E/C/F/TAF
Serious Adverse Events (participants affected / at risk) | 12/112 | 3/58 | 35/273
Other Adverse Events (participants affected / at risk) | 91/112 | 48/58 | 215/273
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E/C/F/TAF (N=112) | E/C/F/TDF (N=58) | All E/C/F/TAF (N=273)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 2
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 2
Appendicitis (Infections and infestations) | 0 | 0 | 4
Cellulitis (Infections and infestations) | 0 | 0 | 2
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Coxsackie viral infection (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus colitis (Infections and infestations) | 1 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 1
Furuncle (Infections and infestations) | 1 | 0 | 1
Hepatitis C (Infections and infestations) | 0 | 0 | 1
Infectious colitis (Infections and infestations) | 0 | 0 | 1
Mycobacterium avium complex infection (Infections and infestations) | 1 | 0 | 1
Neurosyphilis (Infections and infestations) | 1 | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 2
Pyelonephritis (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 1
Viral rash (Infections and infestations) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Vertebral artery dissection (Nervous system disorders) | 0 | 0 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 3
Depression (Psychiatric disorders) | 1 | 2 | 3
Drug abuse (Psychiatric disorders) | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 2 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E/C/F/TAF (N=112) | E/C/F/TDF (N=58) | All E/C/F/TAF (N=273)
Hypogonadism (Endocrine disorders) | 7 | 0 | 12
Constipation (Gastrointestinal disorders) | 4 | 3 | 10
Diarrhoea (Gastrointestinal disorders) | 19 | 9 | 40
Dyspepsia (Gastrointestinal disorders) | 4 | 3 | 9
Flatulence (Gastrointestinal disorders) | 6 | 2 | 6
Nausea (Gastrointestinal disorders) | 25 | 7 | 35
Toothache (Gastrointestinal disorders) | 3 | 1 | 15
Vomiting (Gastrointestinal disorders) | 9 | 4 | 17
Fatigue (General disorders) | 18 | 5 | 29
Seasonal allergy (Immune system disorders) | 4 | 3 | 11
Acarodermatitis (Infections and infestations) | 4 | 3 | 8
Bronchitis (Infections and infestations) | 7 | 3 | 33
Chlamydial infection (Infections and infestations) | 3 | 2 | 16
Conjunctivitis (Infections and infestations) | 9 | 0 | 18
Gastroenteritis (Infections and infestations) | 4 | 2 | 26
Influenza (Infections and infestations) | 8 | 0 | 19
Nasopharyngitis (Infections and infestations) | 7 | 2 | 31
Pharyngitis (Infections and infestations) | 10 | 2 | 20
Sinusitis (Infections and infestations) | 7 | 3 | 28
Syphilis (Infections and infestations) | 5 | 3 | 38
Upper respiratory tract infection (Infections and infestations) | 17 | 12 | 60
Procedural pain (Injury, poisoning and procedural complications) | 3 | 2 | 14
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 | 1 | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2 | 18
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 8 | 27
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 4
Osteopenia (Musculoskeletal and connective tissue disorders) | 4 | 2 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 12
Anorectal human papilloma virus infection (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 4 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 4
Headache (Nervous system disorders) | 11 | 8 | 26
Paraesthesia (Nervous system disorders) | 3 | 4 | 7
Abnormal dreams (Psychiatric disorders) | 8 | 1 | 8
Anxiety (Psychiatric disorders) | 4 | 5 | 15
Depression (Psychiatric disorders) | 11 | 2 | 27
Insomnia (Psychiatric disorders) | 6 | 4 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 6 | 36
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 14
Rash (Skin and subcutaneous tissue disorders) | 11 | 3 | 22

LIMITATIONS AND CAVEATS:
There were no limitations affecting the analysis or results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years